CLINICAL TRIAL: NCT02459574
Title: Ablation Verses Anti-arrhythmic Therapy for Reducing All Hospital Episodes From Recurrent Atrial Fibrillation
Acronym: AVATAR-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AVATAR-AF
Record Dates: First submitted 2015-04-24; First posted 2015-06-02 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure; Recurrent Atrial Fibrillation
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation | interventions — Amiodarone; Sotalol; Adrenergic beta-Antagonists; Calcium Channel Blockers; Flecainide; Propafenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 3-Conventional AF Ablation (Active Comparator): This will involve an ablation procedure carried out in the usual manner. The patient will have three sheaths placed in the leg veins. Catheters will be passed up to the patient's heart from these veins. Two crossing are required into the left atrium. The ablation will involve freeze technology using the Advance Cryoballoon. It will include measuring the electrical signals and may also involve radiofrequency or 'burning' technology in addition.
  Interventions: Procedure: Conventional AF ablation
- Group 2-Anti-arrhythmic therapy (Active Comparator): Anti-arrhythmic drugs: On the treatment start date the patient will have a new tablet prescribed or a change in the dosage of the medication. The patient will be reviewed at 8wks (visit 1) later to see if the medication is working. If the tablets are working, the patients medication will be left unchanged. If not, an alternative tablet or a higher dose will be used.
  Interventions: Drug: Anti-Arrhythmic therapy
- Group 1-AVATAR-AF Ablation Protocol (Experimental): AF ablation with pulmonary vein isolation. The patient will have two sheaths in their leg veins instead of the usual three sheaths. Catheters will be passed up to the heart from these leg veins. The single crossing into the left atrium will be by the usual method. Veins will be ablated using freeze technology known as the Advance Cryoballoon. After the ablation is completed the patient will have scans on their heart and checks of the leg veins. If all the checks are satisfactory at six hours after the procedure the patient will be allowed to go home on the same day. The patient will be reviewed in clinic in 8 weeks (visit 1) after the procedure and if it has been successful, will be reviewed again a month later (visit 2) and if all is well, the patient will be discharged from clinic.
  Interventions: Procedure: AVATAR-AF ablation

INTERVENTIONS:
Procedure: AVATAR-AF ablation — Experimental ablation protocol
  Other Names: Ablation method-surgical
  Arms: Group 1-AVATAR-AF Ablation Protocol
Drug: Anti-Arrhythmic therapy — Group 2 will be prescribed medication listed below:
  Amiodarone; Dronaderone; Sotalol Beta blockers; Calcium channel blockers; Flecainide; or Propafenone.
  You will then be discharged from clinic. A research nurse will contact you by phone to make sure there are no problems and can make hospital appointments if needed.
  Other Names: Amiodarone; Dronaderone; Sotalol; Beta blockers; Calcium channel blockers; Flecainide; Propafenone
  Arms: Group 2-Anti-arrhythmic therapy
Procedure: Conventional AF ablation — Conventional ablation procedure
  Other Names: Ablation method-surgical
  Arms: Group 3-Conventional AF Ablation

SUMMARY:
A streamlined AF ablation procedure done without PV mapping as a daycase is more effective than anti-arrhythmic drugs at reducing all hospital episodes for recurrent atrial fibrillation.

DETAILED DESCRIPTION:
AVATAR-AF is a multicentre, randomised controlled study comparing a streamlined AVATAR-protocol ablation procedure to anti-arrhythmic therapy in patients with documented paroxysmal AF who are considered to be failing current strategy for AF. A secondary control arm will also compare the AVATAR-protocol to conventional AF ablation. 300 patients who are on no prior anti-arrhythmic, 'pill-in-pocket' or taking regular anti-arrhythmics will be randomised in a 1:1:1 manner to a treatment strategy of either AVATAR-protocol ablation, anti-arrhythmic therapy or conventional AF ablation and followed-up for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Documented paroxysmal atrial fibrillation
2. Modification or initiation of anti-arrhythmic agent required for symptom control
3. Males or females eighteen (18) to eighty (80) years of age
4. Suitable candidate for catheter ablation
5. Signed informed consent

Exclusion Criteria:

1. Contraindication to catheter ablation
2. No carer to enable daycase discharge
3. Arrhythmias other than AF documented unless they have had curative ablation (eg. for atrial flutter)
4. No documentation of sinus rhythm within 3 months
5. Valvular or coronary heart disease needing regular follow up
6. EF <45% or moderate/severe LV dysfunction
7. Active gastrointestinal disease
8. Renal failure with creatinine >200 μmol/L or on dialysis
9. Active fever or infection
10. Life expectancy shorter than the trial
11. Allergy to contrast
12. Severe cerebrovascular disease
13. Bleeding or clotting disorders or inability to receive heparin
14. Uncontrolled diabetes (HbA1c ≥73 mmol/mol or HbA1c ≤64 mmol/mol and Fasting Blood Glucose ≥9.2 mmol/L)
15. Serum Potassium [K+] <3.5 mmol/L or >5.0 mmol/L
16. Malignancy needing surgery, chemotherapy or radiotherapy
17. Pregnancy or women of child-bearing potential not using a highly effective method of contraception
18. Must not have previous (4 weeks prior to screening) or current participation in another clinical trial with an investigational drug or investigational device
19. Unable to give informed consent
20. Uncontrolled thyroid disease defined as abnormal thyroid function tests causing cardiac manifestations within the last 6mths
21. Unable to attend follow up visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Prapa Kanagaratnam, Principal Investigator — Imperial College London
Locations (13):
- United Kingdom (13):
  - The Royal Bournemouth Hospital, Bournemouth
  - Brighton University Hospital, Brighton
  - Coventry University Hospital, Coventry
  - Eastbourne District General Hospital, Eastbourne
  - Castle Hill Hospital, Hull
  - Leeds General Infirmary, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - Hammersmith Hospital, London
  - Freeman Hospital, Newcastle
  - Queen Alexandra Hospital, Portsmouth
  - Sheffield University Hospital, Sheffield
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Result] Kanagaratnam P, McCready J, Tayebjee M, Shepherd E, Sasikaran T, Todd D, Johnson N, Kyriacou A, Hayat S, Hobson NA, Mann I, Balasubramaniam R, Whinnett Z, Earley M, Petkar S, Veasey R, Kirubakaran S, Coyle C, Kim MY, Lim PB, O'Neill J, Davies DW, Peters NS, Babalis D, Linton N, Falaschetti E, Tanner M, Shah J, Poulter N. Ablation versus anti-arrhythmic therapy for reducing all hospital episodes from recurrent atrial fibrillation: a prospective, randomized, multi-centre, open label trial. Europace. 2023 Mar 30;25(3):863-872. doi: 10.1093/europace/euac253. PMID 36576323
- [Derived] Mann I, Sasikaran T, Sandler B, Babalis D, Johnson N, Falaschetti E, Copley A, Tayebjee M, Todd D, Shepherd E, McCready J, Poulter N F, Kanagaratnam P. Ablation versus Anti-Arrhythmic Therapy for Reducing All Hospital Episodes from Recurrent Atrial Fibrillation (AVATAR-AF): Design and rationale. Am Heart J. 2019 Aug;214:36-45. doi: 10.1016/j.ahj.2019.04.015. Epub 2019 May 3. PMID 31152874

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2-Anti-arrhythmic Therapy: Anti-arrhythmic drugs: On the treatment start date the patient will have a new tablet prescribed or a change in the dosage of the medication. The patient will be reviewed at 8wks (visit 1) later to see if the medication is working. If the tablets are working, the patients medication will be left unchanged. If not, an alternative tablet or a higher dose will be used.
  Anti-Arrhythmic therapy: Group 2 will be prescribed medication listed below:
  Amiodarone; Dronaderone; Sotalol Beta blockers; Calcium channel blockers; Flecainide; or Propafenone.
  You will then be discharged from clinic. A research nurse will contact you by phone to make sure there are no problems and can make hospital appointments if needed.
Period: Overall Study
Arm/Group | Group 3-Conventional AF Ablation | Group 2-Anti-arrhythmic Therapy | Group 1-AVATAR-AF Ablation Protocol
Started | 108 | 103 | 110
Completed | 101 | 95 | 108
Not Completed | 7 | 8 | 2
Not completed — Withdrawal by Subject | 6 | 6 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Death | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: ITT analysis population (all randomised)
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 3-Conventional AF Ablation | Group 2-Anti-arrhythmic Therapy | Group 1-AVATAR-AF Ablation Protocol | Total
Number analyzed (Participants) | 108 | 103 | 110 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (12.22) | 60.5 (10.34) | 60.1 (9.00) | 60.1 (10.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 46 | 46 | 134
  Male | 66 | 57 | 64 | 187
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Asian | 3 | 1 | 0 | 4
  Ethnicity: Black | 1 | 0 | 0 | 1
  Ethnicity: Chinese | 0 | 1 | 0 | 1
  Ethnicity: Mixed | 0 | 0 | 2 | 2
  Ethnicity: White | 104 | 100 | 108 | 312
  Ethnicity: Other | 0 | 1 | 0 | 1
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m^2] — Population: Missing BMI data for 4nr participants
  kg/m^2
    number analyzed (Participants) | 107 | 100 | 110 | 317
    (all) | 28.88 (4.670) | 27.98 (4.830) | 29.12 (5.040) | 28.68 (4.860)
No. with Hypertension [Count of Participants; unit: Participants]
  Non-Hypertensive | 79 | 67 | 72 | 218
  Hypertensive | 29 | 36 | 38 | 103
CHADSVASc Score (congestive heart failure, hypertension) [Count of Participants; unit: Participants] — The CHADSVASc scoring system assigns 1 point for ages 65-74, 2 points for age ≥75, 1 point for female sex, 1 point for congestive heart failure, 1 point for hypertension, 2 points for history of stroke, transient ischemic attack, or history of thromboembolism, 1 point for vascular disease, and 1 point for Diabetes mellitus.
  The score ranges from 0 to 9 points, and patients are categorized as low risk (score 0), medium risk (score 1), or high risk (score 2 or higher). Population: The full name for CHADSVASc is Congestive Heart Failure, Hypertension, Age ≥75 (Doubled), Diabetes Mellitus, Prior Stroke or Transient Ischemic Attack (Doubled), Vascular Disease, Age 65-74, Sex category.
  CHADSVASc missing for 3nr participants
  Participants
    number analyzed (Participants) | 107 | 102 | 109 | 318
    0 | 43 | 36 | 35 | 114
    1 | 22 | 24 | 30 | 76
    2 | 23 | 19 | 28 | 70
    3 | 10 | 17 | 12 | 39
    4 | 6 | 4 | 4 | 14
    5 | 1 | 1 | 0 | 2
    6 | 2 | 1 | 0 | 3
Ejection Fraction [Mean (Standard Deviation); unit: %] — Population: 44 participants EJF missing at BL
  %
    number analyzed (Participants) | 93 | 93 | 91 | 277
    (all) | 58.3 (5.00) | 57.9 (5.60) | 57.1 (4.88) | 57.8 (5.18)

OUTCOME MEASURES:

1. Primary Outcome: All Hospital Episodes (Emergency Room or Patient Request for OPD) Related to Treatment for Atrial Arrhythmia
Description: Composite outcome measure - Hospital episodes (Emergency Room or Patient Request for OPD) Related to Treatment for Atrial Arrhythmia
Time Frame: 12 months
Population: All randomized participants are eligible for ITT analysis - however, any patients that withdraw prior to first intervention cannot be assessed for the time-to-event based analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3-Conventional AF Ablation | Group 2-Anti-arrhythmic Therapy | Group 1-AVATAR-AF Ablation Protocol
Number analyzed (Participants) | 106 | 100 | 109
Participants | 19 | 76 | 23
Statistical Analysis 1: Comparison: Group 2-Anti-arrhythmic Therapy vs Group 1-AVATAR-AF Ablation Protocol; Primary Analysis - AVATAR-AF vs Anti-Arrhythmic Therapy; Test type: Superiority; p < 0.0001, Log Rank — Bonferonni corrected alpha of 0.05/2 = 0.025; Hazard Ratio (HR) = 0.156, 95% CI 2-sided [0.097 to 0.250] — 95% Wald Confidence Limits Point estimate relates to AVATAR-AF in relation to Anti-Arrhythmic Therapy
Statistical Analysis 2: Comparison: Group 3-Conventional AF Ablation vs Group 1-AVATAR-AF Ablation Protocol; Secondary analysis of Primary Outcome measure - AVATAR-AF vs Conventional Ablation; Test type: Superiority; p = 0.6061, Log Rank — Bonferonni corrected alpha 0.05/2 = 0.025; Hazard Ratio (HR) = 1.173, 95% CI 2-sided [0.639 to 2.154] — 95% Wald Confidence Limits Point estimate relates to AVATAR-AF in relation to Conventional Ablation

2. Secondary Outcome: Death or Stroke From Any Cause
Description: Composite outcome measure
Time Frame: 12 months
Population: Full ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 3-Conventional AF Ablation | Group 2-Anti-arrhythmic Therapy | Group 1-AVATAR-AF Ablation Protocol
Number analyzed (Participants) | 108 | 103 | 110
Participants | 0 | 1 | 0

3. Secondary Outcome: Any Complications Caused by the Procedure (Pericardial Effusion, Bleeding >2 Units, Phrenic Nerve Palsy and Other) or the Anti-arrhythmic Drug (GI Disturbance, Skin Irritation and Other)
Description: Composite outcome measure - Caused by the Procedure (Pericardial Effusion, Bleeding >2 Units, Phrenic Nerve Palsy and Other) or the Anti-arrhythmic Drug (GI Disturbance, Skin Irritation and Other)
Time Frame: 12 months
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Group 3-Conventional AF Ablation | Group 2-Anti-arrhythmic Therapy | Group 1-AVATAR-AF Ablation Protocol
Number analyzed (Participants) | 108 | 103 | 110
participants
  All Events | 3 | 19 | 7
  Drug Side Effect/Allergic Reaction | 1 | 18 | 2
  Vascular Complication | 1 | 0 | 3
  Cardiac Tamponade | 0 | 0 | 2
  Phrenic Nerve Palsy | 0 | 0 | 0
  TIA | 1 | 1 | 0

4. Secondary Outcome: All Hospital Episodes Which Result in a Change in Therapy for Atrial Arrhythmia
Description: Composite outcome measure - All hospital episodes which result in a change in therapy for atrial arrhythmia
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AE's are collected from Randomization up to 1-year end-of-Study Visit
Description: All SAE's were reviewed by an independent Data Monitoring and Safety Board (DSMB)
Arm/Group | Group 3-Conventional AF Ablation | Group 2-Anti-arrhythmic Therapy | Group 1-AVATAR-AF Ablation Protocol
All-Cause Mortality (participants affected / at risk) | 0/108 | 1/103 | 0/110
Serious Adverse Events (participants affected / at risk) | 16/108 | 12/103 | 13/110
Other Adverse Events (participants affected / at risk) | 43/108 | 50/103 | 57/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 3-Conventional AF Ablation (N=108) | Group 2-Anti-arrhythmic Therapy (N=103) | Group 1-AVATAR-AF Ablation Protocol (N=110)
Death (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation/Flutter (Cardiac disorders) | 2 (3) | 5 (5) | 5 (6)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tamponade (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Mass In Left Atrium (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (Cardiac disorders) | 2 (2) | 3 (3) | 1 (1)
Bilateral Papilledema. (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Palpitation (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Right Arm And Face Numbness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Injury To Right Hand (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia & Bronchospasm. (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Nose Surgery (Investigations) | 0 (0) | 1 (1) | 0 (0)
Bleeding From Groin (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pelvic Floor Repair (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fractured Ribs, Cuts And Bruises. (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Strand Of Likely Thrombus Attached To Septum (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hip Replacement. (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Femoral Entry Wound (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Knee Replacement (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
TIA (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 3-Conventional AF Ablation (N=108) | Group 2-Anti-arrhythmic Therapy (N=103) | Group 1-AVATAR-AF Ablation Protocol (N=110)
Atrial Fibrillation (Cardiac disorders) | 6 (7) | 11 (11) | 11 (16)
Palpitations (Cardiac disorders) | 4 (7) | 4 (4) | 6 (6)
All other events < 5% Freq (Investigations) | 33 (57) | 42 (67) | 48 (75)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT02459574/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT02459574/SAP_001.pdf